CLINICAL TRIAL: NCT02350751
Title: A Phase 1 Double-blind, Single-dose, Placebo-controlled, Dose-escalation Study to Evaluate the Safety and Pharmacokinetics of MEDI8852 in Healthy Adults
Brief Title: Phase 1 Placebo-controlled,Dose-escalation Study to Evaluate the Safety and Pharmacokinetics of MEDI8852 in Adults
Acronym: MEDI8852
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D6000C00001
Record Dates: First submitted 2014-12-23; First posted 2015-01-30 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Influenza
Keywords: Influenza, Flu, Flu A, Influenza A
MeSH Terms: conditions — Influenza, Human | interventions — MEDI8852

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MEDI8852 (Experimental): MEDI8852 is a human IgG1 kappa monoclonal antibody (mAb) supplied as 50 mg/mL solution for infusion. MEDI8852 is being evaluated for treatment of patients hospitalized with influenza A.
  Interventions: Drug: MEDI8852
- Placebo (Placebo Comparator): Solution containing no active ingredients
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MEDI8852
  Arms: MEDI8852
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics of MEDI8852 compared to placebo when administered to healthy adult subjects.

DETAILED DESCRIPTION:
This is a phase 1, single-dose, double-blind, placebo-controlled, dose-escalation study to evaluate the safety and pharmacokinetics of MEDI8852 compared to placebo when administered to healthy adult subjects. Approximately 40 subjects will be entered to receive treatment across 4 fixed dose cohorts at 1 site. Investigational product will be delivered intravenously (IV). A total of 4 different dose levels of investigational product will be evaluated across the cohorts. Subjects will be followed for approximately 100 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 through 65 years at the time of screening
2. Weight ≥ 45 kg and ≤ 110 kg at screening
3. Healthy by medical history, physical examination, and baseline safety laboratory studies.
4. Systolic blood pressure (BP) < 140 mm Hg and diastolic BP < 90 mm Hg at screening
5. Electrocardiogram without clinically significant abnormalities at screening
6. Able to complete the follow-up period through Day 101 as required by the protocol
7. Females of childbearing potential who are sexually active with a nonsterilized male partner must use a highly effective method of contraception for at least 28 days prior to the first dose of investigational product and must agree to continue using such precautions through Day 101 of the study

Exclusion Criteria:

1. Acute illness, including fever > 99.5°F, on day prior to or day of planned dosing
2. Any drug therapy within 7 days prior to Day 1 (except contraceptives or a single use of acetaminophen, aspirin, antihistamine. and other nutritional supplements that have not been taken for at least 30 days prior to enrollment, are not exclusionary.
3. Blood drawn in excess of a total of 450 mL (1 unit) for any reason within 2 months prior to screening
4. Receipt of immunoglobulin or blood products within 6 months prior to screening
5. Receipt of any vaccine within 14 days prior to investigational product dosing or planned receipt of any influenza vaccine within 100 days after investigational product dosing
6. Either history of active infection with hepatitis B or C or positive test for hepatitis C or for hepatitis B surface antigen at screening
7. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), or serum creatinine above the upper limit of normal or hemoglobin, white blood cell count, or platelet count below the lower limit of normal at screening
8. History of malignancy other than treated non-melanoma skin cancers or locally-treated cervical cancer in previous 5 years
9. Pregnant or nursing mother
10. History of alcohol or drug abuse within the past 2 years tha OR positive Class A drug screen for amphetamines, barbiturates, opiates, or cocaine at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and tolerability of MEDI8852 | 100 days postdose
  Occurrence of adverse events, serious adverse events, adverse events of special interest, and new onset chronic disease.
Number of Participants with Adverse Events as a Measure of Safety and tolerability of MEDI8852 | 28 days postdose
  Clinical laboratory assessments (ie, serum chemistry, hematology, and urinalysis)

SECONDARY OUTCOMES:
Pharmacokinetics of MEDI8852 in serum: terminal-phase elimination (t½) | 100 days postdose
  This variable will be estimated for MEDI8852 in the IV cohorts where the data allow.
Pharmacokinetics of MEDI8852 in serum: systemic clearance (CL) | 100 days postdose
  This variable will be estimated for MEDI8852 in the IV cohorts where the data allows.
Pharmacokinetics of MEDI8852 in serum: time to maximum serum concentration (Cmax) | 100 days postdose
  This variable will be estimated for MEDI8852 in the IV cohorts where the data allow.
Pharmacokinetics of MEDI8852 in serum: area under the concentration time curve from 0 to t (AUC 0-t) and from 0 to infinity (AUC 0-inf) | 100 days postdose
  This variable will be estimated for MEDI8852 in the IV cohorts where the data allow.
Incidence of anti-drug antibody to MEDI8852 in serum | 100 days postdose
  This variable will be estimated for MEDI8852 in the IV cohorts where the data allow.
Pharmacokinetics of MEDI8852 in serum:volume at steady state (Vss) | 100 days postdose
  This variable will be estimated for MEDI8852 in the IV cohorts where the data allow.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Mallory RM, Ali SO, Takas T, Kankam M, Dubovsky F, Tseng L. A phase 1 study to evaluate the safety and pharmacokinetics of MEDI8852, an anti-influenza A monoclonal antibody, in healthy adult volunteers. Biologicals. 2017 Nov;50:81-86. doi: 10.1016/j.biologicals.2017.08.007. Epub 2017 Aug 23. PMID 28844541